CLINICAL TRIAL: NCT02074813
Title: Effects of Inspiratory Muscle Training (IMT) on Dyspnea in COPD During Pulmonary Rehabilitation: Randomized Controlled Trial
Brief Title: Inspiratory Muscle Training During Pulmonary Rehabilitation in COPD
Acronym: EMI II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMI II (RB 13.124)
Record Dates: First submitted 2014-02-27; First posted 2014-02-28 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Inspiratory muscle training; COPD; dyspnea; Multidimensional Dyspnea Profile questionnaire (MDP).; pulmonary rehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard (No Intervention): conventional pulmonary rehabilitation
- Inspiratory muscle training (Experimental): Inspiratory muscle training associated with a conventional pulmonary rehabilitation
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — Inspiratory muscle training
  Arms: Inspiratory muscle training

SUMMARY:
Demonstrate that IMT associated with a conventional pulmonary rehabilitation program allows a significant improvement of dyspnea in subjects with severe or very severe COPD than a conventional pulmonary rehabilitation program alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD stage 3 or 4
* Hospitalized in the pulmonary rehabilitation unit in the hospital of Morlaix, with a 3 weeks pulmonary rehabilitation course;

Exclusion Criteria:

* FEV ≥ 50%
* Pneumonectomy, Lobectomy less than 6 months
* Patient with risk of spontaneous pneumothorax or rib fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Dyspnea measure | 21 - 4 days / +7 jours
  Measure of dyspnea with the Multidimensional Dyspnea Profile (MDP) questionnaire.

SECONDARY OUTCOMES:
PI max variation | 21 - 4 days / +7 days
  Measure of PI max variation with MicroRPM
CI variation | 21 - 4 days / +7 days
  Measure of CI variation with spirobank II
Dyspnea measure | 21 - 4 days / +7 days
  Meausre of dyspnea with London Chest of Activity Daily Living (LCADL)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre des maladies respiratoires et allergiques - Les Acacias, Briançon, France
  - Brest University Hospital, Morlaix, France

REFERENCES:
- [Derived] Beaumont M, Couasnon C, Peran L, Berriet AC, Ber CL, Pichon R. Determination of the minimal important difference for inspiratory muscle strength in people with severe and very severe COPD. Clin Rehabil. 2023 Nov;37(11):1521-1532. doi: 10.1177/02692155231174124. Epub 2023 May 15. PMID 37186772
- [Derived] Beaumont M, Mialon P, Le Ber C, Le Mevel P, Peran L, Meurisse O, Morelot-Panzini C, Dion A, Couturaud F. Effects of inspiratory muscle training on dyspnoea in severe COPD patients during pulmonary rehabilitation: controlled randomised trial. Eur Respir J. 2018 Jan 25;51(1):1701107. doi: 10.1183/13993003.01107-2017. Print 2018 Jan. PMID 29371379